# Phase II Study of the Combination of Mitoxantrone, Etoposide and Gemtuzumab Ozogamicin (MEGO) for Patients with Acute Myeloid Leukemia Refractory to Initial Standard Induction Therapy

July 25, 2022 Version 5

### PRINCIPAL INVESTIGATOR

Robert Redner, MD

Clinical Instructor, Division of Hematology/Oncology

**UPMC Cancer Pavilion** 

5115 Centre Avenue, 4th

FloorPittsburgh, PA 15232

Phone: 412-864-6625

Email: rednerrl@upmc.edu

### **BIOSTATISTICIAN**

Daniel P. Normolle, PhD

**Biostatistics Facility** 

**UPMC Hillman Cancer Center** 

Suite 325 Sterling Plaza 201

North Craig St.

Pittsburgh, PA 15213

Phone: 412-383-1581

Email: dpn7@pitt.edu

| Т | able of Contents | Page |
|-------|--------------------------------------------|------|
| 1.0 | INTRODUCTION | 4 |
| 4.4 | Charda a bia akina | 4 |
| 1.1 | Study objectives | 4 |
| 1.2 | Background and Rationale | 4 |
| 2.0 | ELIGIBILITY ASSESSMENT AND ENROLLMENT | |
| 2.1 | Eligibility Criteria | 9 |
| 2.2 | Exclusion criteria | 10 |
| 2.3 | Eligibility evaluation | 11 |
| 3.0 | STUDY IMPLEMENTATION | |
| 3.1 | Study design and treatment plan | 12 |
| 3.2 | Off study criteria for the trial | 13 |
| 3.3 | Off treatment criteria for the trial | 13 |
| 4.0 C | ON STUDY EVALUATION | 13 |
| 5.0 | STATISTICAL CONSIDERATIONS AND METHODOLOGY | |
| 5.1 | Number and evaluability of patients | 14 |
| 5.2 | Sample size / Accrual rate | 15 |
| 5.3 | Study Design | 15 |
| 5.4 | Statistical Analysis Plan | 17 |
| 7.0 | ADVERSE EVENT REPORTING | 20 |
| 8.0 | DATA SAFETY MONITORING PLAN | 23 |

| 9.0 STUDY EVALUATION, TREATMENT SCHEMA AND FLOW CHART | 25 |
|-------------------------------------------------------|----|
| 10.0 Drug information | 32 |
| 11.0 References | 40 |

# 1.0 INTRODUCTION

## 1.1 Study objectives

Primary Objective: To evaluate the response rate and toxicity of the combination of mitoxantrone, etoposide and gemtuzumab ozogamicin as second line therapy in patients with acute myeloid leukemia (AML) who have failed the first induction therapy.

Secondary Objectives: To assess the progression-free survival, overall survival and treatment related mortality in patients with AML treated with the combination of mitoxantrone, etoposide and gemtuzumab ozogamicin.

To explore if age, cytogenetic status, percent of blast in the bone marrow prior to therapy or percent expression of CD33 in the leukemia blasts are predictive of complete remission, overall survival or progression-free survival in patients with AML treated with the combination of mitoxantrone, etoposide and gemtuzumab ozogamicin.

## 1.2 Background and Rationale

Acute myeloid leukemia (AML) is a disease characterized by a clonal proliferation of myeloid precursors with reduced capacity to differentiate into more mature cellular elements. As a result, there is an accumulation of leukemic forms in the bone marrow, peripheral blood and other tissues, with a marked reduction in red cells, platelets, and neutrophils. The increased production of malignant cells, along with reduction in these mature elements, results in a

variety of systemic symptoms and signs. These include anemia, bleeding and an increased risk of infection. If left untreated, AML can lead to death within weeks<sup>1</sup>.

The standard treatment for newly diagnosed AML has not changed appreciably over the last few decades and consists primarily of an anthracycline (e.g. daunorubicin, idarubicin) combined with a nucleoside analogue, cytarabine. The goal of remission induction chemotherapy is the rapid restoration of normal bone marrow function<sup>2</sup>. Obtaining complete remission (CR) varies substantially depending on several factors, most notably age and cytogenetic abnormalities at the time of AML diagnosis. CR rates of 65-80% can be expected in younger patients (variably defined as < 55-60 years). CR rates decrease to 30% to 50% in older patients<sup>3</sup>.

There is no agreed standard of care for AML patients that do not respond to initial first line induction therapy. Although remission after second-line therapy may occur, the CR rate is considerably lower. A number of chemotherapy regimens have been used in patients with resistant disease with overall CR rates of 20-40%. These regimens include different combinations and doses of agents that are effective in the treatment of AML such as fludarabine, cytarabine, etoposide, and mitoxantrone<sup>4</sup>.

Gemtuzumab ozogamicin (GO) is an antibody drug conjugate consisting of a recombinant humanized antibody to CD33 which is linked to calicheamicin<sup>5</sup>. Calicheamicin is a potent antitumor antibiotic that cleaves double-stranded DNA at specific sequences<sup>6</sup>. Approximately 90% of AML patients have myeloid blast cells expressing the CD33 surface antigen<sup>7</sup>. Monotherapy with GO resulted in CR of 20-25% in adults with CD33 positive AML in first relapse<sup>8</sup>. GO was approved by the United States Food and Drug Administration (FDA) for use in patients age 60 or older with CD33+ AML in first relapse who were not considered candidates for cytotoxic chemotherapy in 2000<sup>9</sup>. However, due to early deaths in a prospective phase 3 randomized study which incorporated GO in the induction phase in one of the arms (SWOG S0106)<sup>10</sup> the manufacturer withdrew the product from the American market in 2010. The SWOG S0106 study used 6 mg/m<sup>2</sup> of GO on day 4 of induction with cytarabine, daunorubicin. The treatment-related mortality (TRM) was 5% on the GO arm vs 1% on the other arm. In 2017, FDA again approved GO for induction therapy in combination with chemotherapy based on a phase 3 prospective randomized, open-label study (ALFA-0701 trial<sup>11</sup>) and as monotherapy for patients unfit for intensive treatment based on the phase 3

randomized EORTC-GIMEMA AML-19 trial<sup>12</sup>. The ALFA-0701 trial randomized 280 patients 50-70 year-old to receive induction with daunorubicin and cytarabine or daunorubicin, cytarabine and GO 3mg/m² on days 1,4,7 of induction. It showed that the addition of GO to the induction chemotherapy improved event-free survival. The AML-19 trial randomized 237 patients unfit for induction chemotherapy to receive either best supportive care or GO 6mg/m² on day 1 and 3mg/m² on day 8. It showed that GO improved the overall survival in patients unfit for intensive treatment when compared to best supportive care with no difference in the adverse events. The NCRI AML17 trial<sup>13</sup> studied further the dose of GO with induction chemotherapy showing that 3mg/m² has the same efficacy but better safety profile than 6mg/m². The dosing regimen of GO as it is currently approved by the US FDA is 3mg/m² (maximum dose 4.5mg) on days 1,4,7 with induction chemotherapy or 6mg/m² on day 1 followed by 3mg/m² on day 8 if used as monotherapy.

The most important GO-associated hematologic toxicity is myelosuppression (thrombocytopenia, neutropenia). Infusion-related adverse reactions are similar to those of other monoclonal antibodies (fever, chills, cutaneous rash, hypotension, hypertension, dyspnea, nausea, emesis and headache). They are usually transient and respond well to symptomatic therapy<sup>14</sup>.

Hepatic veno-occlusive disease or sinusoidal obstructive syndrome (VOD/SOS) is the most frequently reported life-threatening non-hematological adverse event. Overall, among all adult GO- treated AML patients evaluated in the clinical trial setting, SOS occurred at a rate of 3% when GO was administered as monotherapy at the initial FDA approved dose and schedule (for relapsed AML, 9 mg/m² on day 1 and 14); 7% when the drug was used in conjunction with other chemotherapeutic agents that are not known to be hepatotoxic; and 28% when GO was combined with thioguanine, a hepatotoxic chemotherapeutic agent. SOS rates were between 15% and 40% if stem cell transplantation was performed within 3 months of GO administration<sup>15</sup>. Another observational study showed an overall 9.1% risk of SOS with GO and 2.7% risk of death from SOS<sup>16</sup>. During the early 2000s when GO was used at higher doses it was observed that patients that received GO <3.5 months before allogeneic stem cell transplantation had much higher incidence of SOS<sup>17</sup>, which was no longer observed in the modern era of lower GO fractionated doses<sup>18</sup>.

Various clinical trials have evaluated the efficacy of GO as monotherapy in newly-diagnosed AML, refractory/relapsed AML and in combination with chemotherapy for induction. Different dosing schedules of GO were used in these trials. In addition to grade 3/4 neutropenia and thrombocytopenia some patients also develop transaminitis and VOD (Table 1).

Table 1: Clinical trials with gemtuzumab ozogamicin

| | No. of | | GO Dosing | Therapy | Results | Ref |
|---|---|---|---|---|---|---|
| | pts | disease | | | | Kei |
| EORTC-<br>GIMEMA<br>AML-19 | 237 | New diagnosis,<br>unwilling or unfit<br>for treatment | Induction: 6 mg/m <sup>2</sup> on day 1 and 3 mg/m <sup>2</sup> on day 8. Maintenance: 2mg/m <sup>2</sup> monthly up to 8 doses | Best<br>Supportive<br>Care<br>GO +/- | CR/CRi 27% on the GO arm. OS improvement at 1 year with GO (4.9 vs 3.6 months, p=0.005) | 12 |
| LRF AML<br>14<br>and<br>NCRI<br>AML 16 | 495 | New diagnosis,<br>unfit for intensive<br>treatment | 5 mg (fixed dose) on<br>day 1 of 42-day<br>cycles for a<br>maximum of four<br>cycles | LDAC 20mg<br>BID on days<br>1-10 of<br>42-day cycles<br>+/-<br>GO | Improved CR with GO (21% vs 11%, P= .002). No difference in OS. Patients in the GO arm had more nausea and vomiting, required more platelet transfusions and longer duration of antibiotics. No episodes of VOD were reported. | 19 |
| MRC<br>AML-15 | 1113 | New diagnosis | 3mg/m² on the first day of induction. | DA or DAE or<br>FLAG-IDA<br>+/-<br>GO | No difference is OS but improved 5-year OS in patients with favorable cytogenetics. No excess hematologic or liver toxicity on the GO arm | 20 |
| ALFA-0701 | 278 | New diagnosis | Induction: 3mg/m² on days 1,4,7 Consolidation: 3mg/m² on day 1 for up to two cycles | Induction<br>DA +/- GO<br>Consolidation:<br>DA +/- GO | Improved EFS, DFS on the intervention arm but no difference in OS. Prolonged thrombocytopenia and neutropenia on the GO arm.3 cases of VOD were reported on the GO arm. | 11,21 |
| NCRI<br>AML16 | 1115 | New diagnosis | Induction: 3 mg/m²<br>on day 1 | DA +/- GO | Improved OS on the treatment arm and similar TRM | 22 |
| SWOG<br>S0106 | 595 | New diagnosis | Induction 6 mg/m²<br>on day 4 | DA (with D at<br>60 mg/m2) vs<br>DA (with D at<br>45mg/m2) plus GO | No difference in OS with increased TRM in the GO arm (6% vs 1%) | 10 |

| EORTC-<br>GIMEMA<br>AML-17 | 472 | New diagnosis | Induction: 6mg/m²<br>on days 1 and 15 | MEC +/- GO | Similar CR rate and OS. Higher TRM with GO (22% vs 18%) mainly driven by patients >70 years old | 23 |
|---|---|---|---|---|---|---|
| | 788 | New diagnosis | Induction: | Randomi- zation | No difference in OS. | |
| NCRI | | | randomization To 3 or | | Increased TRM with higher | 13 |
| | | | 6 mg/m <sup>2</sup> | | | |
| AML17 | | | on day 1 | to ADE or DA, | GO dose. | |
| | | | | both + GO | | |
| HOVON-43 | 232 | Consolidation | 6 mg/m <sup>2</sup> every 4 | | No difference in OS | 24 |
| | | | weeks, up to 3 cycles | Observation vs GO | | Z+ |

**Abbreviations:** CR, complete remission; CRi, complete remission with incomplete hematologic recovery; GO, Gemtuzumab Ozogamicin; OS, overall survival; LDAC, low-dose cytarabine; VOD, veno-occlusive disease, DA, daunorubicin + cytarabine, DAE, daunorubicin + cytarabine + etoposide; FLAG-IDA, fludarabine + cytarabine + G-CSF + idarubicin; EFS, event-free survival; DFS, disease-free survival; TRM, treatment-related mortality; MEC, mitoxantrone + etoposide + cytarabine; ADE, cytarabine + daunarubicin + etoposide

## **Rationale**

The combination of mitoxantrone and etoposide is an active regimen in refractory/relapsed AML patients<sup>25</sup>. In a retrospective study, we evaluated the efficacy and toxicity of mitoxantrone and etoposide in AML patients treated at our institution who did not respond to first induction therapy with cytarabine and an anthracycline. A total of thirty-five AML patients were treated with mitoxantrone (10 mg/m²/d) on days 1-5 and etoposide (100 mg/m²/d) on days 1-5. Thirteen of thirty-five patients (37%) achieved CR. There were no grade 3/4 hepatic toxicities. The median duration of neutropenia in patients achieving CR was 29 days after reinduction. 14% of patients died from infectious complications.

In order to increase the efficacy of mitoxantrone and etoposide as second line therapy in patients with AML we propose to conduct a phase II clinical trial evaluating the safety and efficacy of the combination of GO, mitoxantrone and etoposide. A similar trial was open in our institution before Pfizer withdrew the drug from the market in 2010<sup>26</sup>. Before the withdrawal 5 patients were treated with a regimen consisted of mitoxantrone 10 mg/m2 administered intravenously on days 1–3, etoposide 100 mg/m2 administered on days 1–5 and on day 6 GO 3 mg/m2. Three of the five patients achieved a CR. There were no treatment-related deaths. All patients developed grade 3–4 neutropenia and thrombocytopenia, with complete responders requiring a median of 19 days (range, 17–34 days) from the completion of

treatment to recover their neutrophils and a median of 24 days (range, 17–34 days) to recover their platelets. One patient developed grade 3 ALT transaminitis that resolved within 24 h and one patient developed a transient ischemic attack. No patient developed clinical signs or symptoms of veno-occlusive disease.

It has been demonstrated that high peripheral CD33-antigen load is an independent adverse prognostic factor in AML patients treated with GO. Data indicate that a high peripheral CD33antigen load consumes a large portion of the GO, which results in reduced GO penetration into the bone marrow <sup>27</sup>. As a consequence, CD33 saturation of AML blast cells present in the bone marrow is incomplete, which may hamper subsequent cell kill. Administration of GO may be more effective after reduction of the leukemic cell burden with conventional chemotherapy. Thus, we plan to administer the GO after the administration of mitoxantrone and etoposide. Furthermore, since enrolled patients in the study will already be treated with combination of cytarabine and an anthracycline (1st regimen) and mitoxantrone and etoposide (2nd regimen) and GO has been associated with neutropenia and thrombocytopenia, we plan to use a single dose of GO 3 mg/m² the day after the completion of the 5 days of etoposide and mitoxantrone.

# 2.0 ELIGIBILITY ASSESSMENT AND ENROLLMENT

#### 2.1 Eligibility Criteria

- 1. Able to understand and have the ability to provide written consent.
- 2. Age:  $\geq$ 18 and  $\leq$ 75 years old.
- 3. Patients with newly diagnosed AML based on the World Health Organization classification who have persistent disease after their first course treatment with an anthracycline and cytarabine (the diagnosis of persistent disease, which is defined as ≥10% blasts by morphology for this trial or >5% blasts if they have had an increase in blasts from the last bone marrow biopsy, will be based on their assessment after bone marrow aspiration and/or biopsy after initial treatment). The bone marrow aspiration and/or biopsy will be evaluated by the Hematopathology Division of the University of Pittsburgh. In order to prevent any delays in starting therapy for eligible patients, a preliminary evaluation of the bone marrow will be sent by the hematopathologist via e-mail to the investigator.

- 4. Patients with myelodysplastic syndrome (MDS) based on the World Health Organization classification who have persistent disease after their treatment with an anthracycline and cytarabine (the diagnosis of persistent disease, which is defined as ≥10% blasts by morphology for this trial or >5% blasts if they have had an increase in blasts from the last bone marrow biopsy, will be based on their assessment after bone marrow aspiration and/or biopsy after initial treatment).
- 5. CD33 expression in ≥ 30% of leukemic blasts on the bone marrow.
- 6. Eastern Cooperative Oncology Group Performance Status of 0 -2 (see Appendix I).
- 7. Patients must have the following laboratory values prior to beginning protocol treatment:
  - Calculated creatinine clearance ≥ 30 mL/min (using the Cockcroft-Gault equation CL creatinine = ((140-age) x body mass X 0.85 if female)/72 x creatinine where age is given in years, body mass is given in Kg and creatinine is given in mg/dl).
  - Aspartate aminotransferase (AST) ≤ 2.5 x upper normal limit.
  - Alanine aminotransferase (ALT) ≤ 2.5 x upper normal limit.
  - Total bilirubin ≤ 2 x upper normal limit.

**Note:** As many eligible patients will be pancytopenic secondary to their disease or prior treatments, hematologic abnormalities will not be used as criteria for entry or exclusion.

- 8. Left ventricular ejection fraction (LVEF) ≥50 %.
- 9. Females of child-bearing potential must have a negative pregnancy test during screening and all subjects must agree to use an effective method of contraception. A woman is eligible to enter and participate in the study if she is of:
  - a. Non-childbearing potential (*i.e.*, physiologically incapable of becoming pregnant) including any female who has had a hysterectomy or has had a bilateral oophorectomy (ovariectomy).
  - b. Childbearing potential, has a negative serum pregnancy test during the screening period and agrees to avoid sexual activity or use contraception from screening through follow-up (method of birth control if the patient is not neutropenic include the use of a diaphragm, intrauterine device, contraceptive sponge and/or usage of male condom with a spermicide from the partner). A man with a female partner of childbearing potential is eligible to enter and participate in the study if he has either had a prior vasectomy or agrees to avoid sexual activity or use adequate contraception (as described above) from screening through follow-up.

#### 2.2 Exclusion criteria

- 1. Patients with a diagnosis of Acute Promyelocytic Leukemia (APL) as defined by the World Health Organization.
- 2. Relapsed acute leukemia.
- 3. Bi-lineage or bi-phenotypic leukemia.
- 4. Prior use of mitoxantrone or etoposide or GO.
- 5. Previous allogeneic hematopoietic cell transplantation.
- 6. First induction course of acute myeloid leukemia with CPX-351.
- 7. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of treating investigator.
- 8. Has known history of active Hepatitis B (HBsAg reactive) or Hepatitis C (detectable HCV RNA).
- 9. Uncontrolled, life-threatening infection that is not responding to antimicrobial therapy.
- 10. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
- 11. Patient may have not received any other investigational anti-neoplastic agents within 4 weeks from the start of therapy.
- 12. Concurrent active malignancy; exceptions include patients who have been disease free for 5 years, patients with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma, or patients with another malignancy with better prognosis than AML.
- 13. Women who are pregnant or breastfeeding.
- 14. Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory or cardiac disease).

#### 2.3 Eligibility evaluation

The following clinical and laboratory assessments must be performed for all eligible patients within 14 days of study enrollment and consent:

- 1. Complete medical history and physical examination, including height, weight, body surface area (BSA), ECOG performance status, and a neurological evaluation.
- 2. Echocardiogram to evaluate cardiac ejection fraction.
- 3. CBC with differential and platelets.
- 4. Complete metabolic panel (Na, K, Cl, CO2, glucose, BUN, Cr, Ca, total protein, albumin, total bilirubin, AST, ALT, and alkaline phosphatase) and magnesium level.
- 5. LDH, uric acid, and phosphorus levels.
- 6. PT/INR, PTT.
- 7. Urinalysis.
- 8. PA and lateral chest x-ray. If clinically indicated CT Chest/Abdomen/Pelvis can be performed.
- 9. EKG.
- 10. Urine pregnancy test for all women  $\leq$  60 years old.

The following clinical and laboratory assessments must have been performed for all eligible patients within 12 weeks from initiation of treatment:

- 1. Hepatitis B surface antigen.
- 2. Hepatitis C antibody and if positive HCV RNA.

#### 3.0 STUDY IMPLEMENTATION

# 3.1 Study design and treatment plan

This study is an open-label, single arm phase II study which will examine the efficacy and toxicity of the combination therapy of GO, mitoxantrone and etoposide in patients who did not respond to first line induction therapy.

#### Treatment plan

Eligible patients will be treated at the UPMC Hillman Cancer Center inpatient leukemia service. Patients will receive mitoxantrone 10mg/m<sup>2</sup> administered intravenous piggyback

(IVPB) in 50ml 0.9% normal saline over 15 minutes on days 1-5 and etoposide 100 mg/m<sup>2</sup> administered intravenously in 500 ml of 0.9% sodium chloride over 2 hours on days 1-5.

On day 6, patients will receive a single dose of GO 3mg/m² (maximum dose 4.5mg). Patients will be pre-medicated 1 hour prior to the GO infusion with diphenhydramine 50mg administered orally or intravenously, acetaminophen 650 mg administered orally or intravenously and 1mg/kg methylprednisolone or an equivalent dose of alternative corticosteroid administered IV within 30 minutes prior to infusion of GO. GO will be administered intravenously in 50 ml (or other suitable volume resulting in a final GO concentration between 0.075 mg/mL to 0.234 mg/mL) of 0.9% sodium chloride over 2 hours. Doses of GO will be based on BSA calculated using actual body weight with a cap of 4.5mg. Vital signs will be recorded within one hour prior to the infusion and then every 30 minutes during the infusion and 30 minutes and one hour after completion of infusion. An additional dose of methylprednisolone 1 mg/kg IV may be given for any sign of infusion reaction, such as fever, chills, hypotension, or dyspnea occurring during the GO infusion or within 4 hours after the GO infusion.

For dose modifications based on kidney and liver function please see the treatment schema at the end of the study.

Supportive care including blood product transfusions, antiemetic medications, antiviral and antifungal medications, growth factor support, tumor lysis syndrome prophylaxis, or empiric antibiotics may be used at the clinical discretion of the provider.

# 3.2 Off study criteria for the study

- 1. Request by the patient at any time for any reason.
- 2. The patient may at any time be removed from the trial at the principal investigator's discretion if the principal investigator deems the patient to be at unacceptable risk to remain on the study. Reasons for this action may include (but are not limited to) diseaseprogression with declining organ function/performance status before treatment; inadequate family/caregiver support; noncompliance.

#### 3.3 Off treatment criteria for the study

- 1. Unacceptable adverse event(s) due to the infusion of any of the three antineoplastic agents which necessitates the termination of the therapy.
- 2. Intercurrent disease that prevents the administration of treatment.

#### 4.0 ON STUDY EVALUATION

All patients enrolled in the study will have the following evaluations:

- History and physical examination will be performed daily during the hospital stay and then weekly (± 4 days) as an outpatient for 4 weeks after discharge and then every 2 weeks until count recovery (defined as ANC ≥1000 with or without PLT ≥ 100,000). Daily weight will be measured (if clinically possible) while in the hospital and at each outpatient visit.
- 2. If patients develop grade 3 or 4 non-hematologic toxicity during their treatment, they will be followed weekly after discharge until resolution of toxicity or improvement to grade 2 or less.
- 3. CBC with differential, complete metabolic panel (Na, K, Cl, CO2, glucose, BUN, Cr, Ca, total protein, albumin, total bilirubin, AST, ALT, and alkaline phosphatase), phosphorus, uric acid, magnesium level and LDH will be performed daily while in the hospital. After discharge, CBC with differential and complete metabolic panel as defined above will be obtained weekly (± 4 days) until count recovery (defined as ANC ≥1000 with or without PLT ≥ 100,000).
- 4. Bone marrow biopsy and/or aspirate will be performed no earlier than 7 days after the therapy completion to evaluate disease response.
- 5. Bone marrow biopsy/aspiration to test for remission will be performed once hematopoietic recovery (defined as ANC ≥1000 with or without PLT ≥ 100,000) has been achieved. It can be performed in the inpatient or outpatient setting. If the bone marrow is consistent with morphologic complete remission, minimal residual disease testing will be performed with flow cytometry. If, on diagnosis, the NPM1 mutation was detectable by PCR or next-generation sequencing, then NPM1 PCR will be performed as well if morphologic complete remission is achieved. If hematopoietic recovery has not been achieved by 5 weeks (± 7 days) after the completion of therapy, bone marrow biopsy and/or aspiration for disease evaluation will be

- performed. If there is no evidence of leukemia, subsequent bone marrow biopsies will be performed based on count recovery.
- 6. After the assessment of the recovery marrow patients will be followed remotely from chart review to evaluate the disease-free survival and the overall survival. If information cannot be obtained from the chart patients may be contacted by telephone.

#### 5.0 STATISTICAL CONSIDERATIONS AND METHODOLOGY

# 5.1 Number and evaluability of patients

This is a phase II study of the combination therapy of GO, mitoxantrone and etoposide as second line therapy in patients with acute myeloid leukemia. The study is designed to assess the therapeutic efficacy and the toxicity profile using Simon's optimal two-stage phase II design to permit early stopping of the trial if there is strong evidence that the studied treatment is inefficacious.

To be evaluable for clinical response, a patient must:

- 1. Receive a total of 5 days of mitoxantrone and etoposide,
- 2. Receive 1 dose of GO and
- 3. Have a follow-up bone marrow biopsy to evaluate the response to therapy.

Additional participants will be recruited to replace those who are not evaluable for clinical response. The accrual target is a maximum of 44 response-evaluable patients. All participants who begin treatment will be counted in the interim analysis for excess mortality.

# 5.2. Sample Size/Accrual rate

#### 5.2.1 Sample size

This study is expected to require a minimum of 16 patients (at the interim evaluation of response) and a maximum of 44 response-evaluable patients unless undue toxicity is encountered. We anticipate accruing up to 9 additional patients (~20%) to account for patients who may prove unevaluable (i.e. ineligibility, cancellations, death or major violations). Therefore, our overall sample size will be a maximum of 53 patients.

#### 5.2.2. Accrual time and study duration

Based on previous efforts in recruiting patients at the UPMC Hillman Cancer Center, it is anticipated that at least thirty patients per year will be enrolled in the protocol and the accrual will be completed within two years. The final evaluation of the study to assess overall survival will be conducted at 5 years or if all subjects expire, whichever comes first.

#### 5.3. Study design

**5.3.1 Definition of complete remission (CR):** An evaluable patient will be classified as having complete remission if they meet the criteria in Appendix II.

<u>Decision Rule (Simon two-stage design):</u> The largest CR rate where the proposed treatment regimen would be considered ineffective in this population is 35%. Subsequent studies will be warranted if the CR rate is 50% or higher or the CR rates are similar to historical data but

the disease-free survival and the overall survival are improved in comparison to our institution's historical cohort. The following optimal Simon two stage design uses 44 patients to test the null hypothesis that the true CR rate in the given patient population is at most 35%.

Stage 1: Enter 16 evaluable patients. If 5 or fewer patients have a CR in this timeframe, we will consider this early evidence that this treatment regimen is not sufficiently efficacious in this patient population, and the accrual of patients will be stopped. If 6 or more patients have a CR, then accrual will continue in the second stage of this trial.

Stage 2: Enter an additional 28 evaluable patients to the trial. If 19 or more patients achievea complete remission, the treatment will be promoted for further consideration. This design has  $\alpha$ =0.15 and  $\beta$ =0.20; the large value of  $\alpha$  is appropriate in an early phase trial. If the probability of CR is 35%, the expected sample size is 30.3 patients, i.e., the probability that the trial will be halted after 16 patients is 48.9%.

### **5.3.2 Monitoring for treatment-induced mortality**

The trial will be continually monitored to ensure that treatment-induced mortality is not excessive, defined as >0.20 of patients treated. A safety-evaluable patient is a patient

who was consented and started the protocol chemotherapy. All safety-evaluable patients, not just those evaluable for clinical response, are counted in the interim analysis for mortality. The cutpoints are listed in Table 2.

**Table 2.** Stopping rule for excessive mortality. The trial will be halted if, for the number of patients in the following table, the number of deaths is greater than or equal to the given number.

| # Patients | # Deaths | # Patients | # Deaths |
|------------|----------|------------|----------|
| 4 | 3 | 24 | 7 |
| 6 | 3 | 26 | 8 |
| 8 | 3 | 28 | 8 |
| 10 | 4 | 30 | 8 |
| 12 | 4 | 32 | 9 |
| 14 | 5 | 34 | 9 |
| 16 | 5 | 36 | 10 |
| 18 | 6 | 38 | 10 |
| 20 | 6 | 40 | 11 |
| 22 | 7 | 42 | 11 |

Justification of the stopping rule: It was assumed that under standard of care, the probability of death is  $\pi$ =0.2. A beta-binomial model is assumed with  $\alpha$ =2 and  $\beta$ =8. If the number of deaths, x, is greater than the value in the Stopping Rule table for the number of patients, n, then:

$$P(\pi > 0.2 | \alpha, \beta, x, n) > 0.75.$$

Under different assumptions of the true probability of death (True P(Death)), the expected number of patients (E(n)) and the probability of the trial stopping early (P(Stop Early)) were determined by Monte Carlo simulation:

| True P(Death) | E(n) | P(Stop Early) |
|---------------|------|---------------|
| 0.20 | 28.3 | 0.513 |
| 0.25 | 22.9 | 0.720 |
| 0.30 | 15.8 | 0.900 |
| 0.35 | 11.5 | 0.973 |
| 0.40 | 8.4 | 0.994 |
| 0.45 | 6.9 | 0.996 |

### 5.4. Statistical analysis plan

#### 5.4.1. Analysis of complete remission

The probability of complete remission (CR, Appendix II) will be estimated by the number of CR divided by the total number of patients evaluable for response. A 95% one-sided exact binomial confidence interval of the form ( $\pi_L$ ,1) for the true probability of CR will be calculated.

#### 5.4.2 Analysis of secondary endpoints

Overall and progression-free survival functions will be estimated by the product limit (Kaplan-Meier) method. The median survival and its 90% confidence interval will also be reported.

Proportional hazards (Cox) regression will be used to describe the relationship between age, cytogenetic status (poor, intermediate, favorable), percent of blast in the bone marrow prior to therapy and percent expression of CD33 in the leukemia blasts to overall and progression-free survival. Likelihood ratio tests will be used to identify statistically significant ratios and profile likelihood confidence intervals will be estimated for hazard ratios of statistically significant predictors. Logistic regression will be applied in a similar fashion to determine predictors of complete remission.

#### 6. ADVERSE EVENT REPORTING

**Definitions** 

The following definitions of terms apply to this section:

<u>Adverse event</u>: Any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.

<u>Life-threatening adverse event or life-threatening suspected adverse reaction</u>: An adverse event or suspected adverse reaction is considered "life-threatening" if, in the view of either the investigator or sponsor, its occurrence places the patient or subject at immediate risk of death. It does not include an adverse event or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

Serious adverse event or serious suspected adverse reaction: An adverse event or

suspected adverse reaction is considered "serious" if, in the view of either the investigator or sponsor, it results in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect. Important medical events that may not result in death,

be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.

<u>Suspected adverse reaction</u>: Any adverse event for which there is a reasonable possibility that the drug caused the adverse event. Suspected adverse reaction implies a lesser degree of certainty about causality than adverse reaction, which means any adverse event caused by a drug.

Adverse reaction means any adverse event caused by a drug. Adverse reactions are a subset of all suspected adverse reactions where there is reason to conclude that the drug caused the event.

<u>Unexpected adverse event or unexpected suspected adverse reaction</u>: An adverse event or suspected adverse reaction is considered "unexpected" if it is not listed in the investigator brochure or is not listed at the specificity or severity that has been observed; or, if an investigator brochure is not required or available, is not consistent with the risk information described in the general investigational plan or elsewhere in the current application, as amended. For example, under this definition, hepatic necrosis would be unexpected (by virtue of greater severity) if the investigator brochure referred only to elevated hepatic enzymes or hepatitis. Similarly, cerebral thromboembolism and cerebral vasculitis would be unexpected (by virtue of greater specificity) if the investigator brochure listed only cerebral vascular accidents. "Unexpected," as used in this definition, also refers to adverse events or suspected adverse reactions that are mentioned in the investigator brochure as occurring with a class of drugs or as anticipated from the pharmacological properties of the drug, but are not specifically mentioned as occurring with the particular drug under investigation.

Eliciting AE Information

Research subjects will be routinely questioned about AEs at study visits.

Recording Requirements

All observed or volunteered adverse events (serious or non-serious) and abnormal test findings, regardless of study group or suspected causal relationship to the study drug(s) will be recorded in the subjects' case histories. For all adverse events, sufficient information will be pursued and/or obtained so as to permit 1) an adequate determination of the outcome of the event (i.e., whether the event should be classified as a *serious adverse event*) and; 2) an assessment of the casual relationship between the adverse event and the study drug(s).

AEs or abnormal test findings felt to be associated with the investigational drug or study treatment(s) will be followed until the event (or its sequelae) or the abnormal test finding resolves or stabilizes at a level acceptable to the Sponsor-Investigator.

# **Abnormal Test Findings**

An abnormal test finding will be classified as an *adverse event* if one or more of the following criteria are met:

- The test finding is accompanied by clinical symptoms.
- The test finding necessitates additional diagnostic evaluation(s) or medical/surgical intervention; including significant additional concomitant drug treatment or other therapy.

**Note**: simply repeating a test finding, in the absence of any of the other listed criteria, does not constitute an AE.

 The test finding leads to a change in study dosing or discontinuation of subject participation in the clinical study.

#### REPORTING OF SERIOUS ADVERSE EVENTS

All events meeting the definition of a serious adverse event, from the date of first dose of study drug until 30 days after last dose, should be reported according to the departmental SAE checklist and SAE form. The initial SAE form should be sent to the following within 24 business hours / 1 business day of the Principal Investigator becoming aware:

- 1. Robert Redner, MD
- 2. CRSSafetySubmissions@upmc.edu
- 3. Local Institutional Review Board when reporting requirements are met.
- 4. Pfizer Safety @ SAEFaxmailbox@Pfizer.com

In addition to completing appropriate patient demographic and suspect medication information, the report should include as applicable the following information that is available at the time of report within the Sections B and C of the departmental SAE form:

- CTCAE(5.0) term(s) and grade(s)
- current status of study drug
- all interventions to address the AE (testing and result, treatment and response)
- hospitalization and/or discharge dates
- event relationship to study drug

# Follow-up reports:

Additional information may be added to a previously submitted report by adding to the original departmental SAE form and submitting it as follow-up or creating supplemental summary information and submitting it as follow-up with the original departmental SAE form. Special Interest Serious Adverse Events

The following events also require reporting to Pfizer at the fax number provided above.

- 1. Exposure during Pregnancy, Exposure during Lactation, Occupational Exposure, and Lack of Effect. Even though there may not be an associated SAE, exposure to the Pfizer drug product during pregnancy, exposure to the Pfizer drug product during lactation, and occupational exposure to the Pfizer drug product are reportable, and lack of effect od rh Pfizer drug product may also be reportable. The term SAE is understood to include exposure during pregnancy, exposure during lactation, occupational exposure, and reportable instances of lack of effect.
- 2. <u>Hy's Law Cases</u>. Cases of potential drug-induced liver injury as assessed by laboratory test values are reportable. If a Subject develops abnormal lab values in aspartate transaminase (AST) or alanine transaminase (ALT) or both, concurrent with abnormal elevations in total bilirubin and no other known cause of liver injury, that event would be classified as a Hy's Law Case. The term SAE is understood to include Hy's Law Cases.

#### 7. DATA SAFETY MONITORING PLAN

Investigator/Sub-investigators, regulatory, CRS management, clinical research coordinators, clinical research associates, data managers, and clinic staff meet regularly in the disease center Data Safety Monitoring Board (DSMB) to review and discuss study data to include, but not limited to, the following:

- · serious adverse events
- subject safety issues
- · recruitment issues
- accrual
- protocol deviations
- unanticipated problems
- breaches of confidentiality

Minutes from the disease center DSMB meetings are available to those who are unable to attend in person.

All toxicities encountered during the study will be evaluated on an ongoing basis according to the NCI Common Toxicity Criteria Version 5.0. All study treatment associated adverse events that are serious, at least possibly related and unexpected will be reported to the IRB. Any modifications necessary to ensure subject safety and decisions to continue or close the trial to accrual are also discussed during these meetings. If any literature becomes available which changes the risk/benefit ratio or suggests that conducting the trial is no longer ethical, the IRB will be notified in the form of an Unanticipated Problem submission and the study may be terminated.

All study data reviewed and discussed during these meetings will be kept confidential. Any breach in subject confidentiality will be reported to the IRB in the form of an Unanticipated Problem submission. The summaries of these meetings are forwarded to the UPMC Hillman Cancer Center DSMC which also meets monthly following a designated format.

For all research protocols, there will be a commitment to comply with the IRB's policies for reporting unanticipated problems involving risk to subjects or others (including adverse events). DSMC progress reports, to include a summary of all serious adverse events and modifications, and approval will be submitted to the IRB at the time of renewal.

Protocols with subjects in long-term (survival) follow-up or protocols in data analysis only, will be reviewed bi-annually.

Both the UPMC Hillman Cancer Center DSMC as well as the individual disease center DSMB have the authority to suspend accrual or further investigate treatment on any trial based on information discussed at these meetings.

All records related to this research study will be stored in a locked environment. Only the researchers affiliated with the research study and their staff will have access to the research records.

# 8. STUDY EVALUATION, TREATMENT SCHEMA AND FLOW CHART

| Pre-treatment evaluation | |
|-------------------------------------------------------|---------------------|
| | Within last 6 weeks |
| | from |
| | day of consent |
| Anti-Hepatitis C antibody and if positive HCV RNA PCR | Х |

| Hepatitis B surface antigen | X |
|---|---|
| | Within 14 days from day of consent |
| Medical history and physical examination | X |
| Height, weight, BSA, ECOG performance status | X |
| Toxicities from prior therapies | X |
| Cardiac echocardiogram | X |
| Bone marrow biopsy and aspiration | X |
| Urine βHCG in women ≤ 60 years old (pregnancy test) | X |
| PT/INR, PTT | X |
| Complete metabolic panel (Na, K, Cl, CO2, glucose, BUN, Cr, Ca, total protein, albumin, total bilirubin, AST, ALT and alkaline phosphatase) | Х |
| Magnesium, Phosphorous, Uric Acid, LDH | X |
| CBC with differential | X |
| Urinalysis | X |
| Electrocardiogram (12 lead) | X |
| Chest radiograph | X |
| CT Chest, Abdomen and/or Pelvis if indicated | X |

| Treatment Schema | | | | | | |
|-----------------------------|-------|-------|-------|-------|-------|-------|
| | Day 1 | Day 2 | Day 3 | Day 4 | Day 5 | Day 6 |
| Mitoxantrone | Х | Х | Х | Х | Х | |
| Etoposide * | Х | Х | Х | Х | Х | |
| Gemtuzumab<br>ozogamicin ** | | | | | | X |

<sup>\*</sup> Dose modification of etoposide for patients who develop elevated total bilirubin and/or AST or decrease in creatinine clearance

| Adverse event | Dose modification of etoposide |
|---|---|
| CrCl 10 – 50 ml/min | administer 75% of normal dose |
| CrCl < 10 ml/min | |
| | administer 50% of normal dose |
| CrCl <50 ml/min | Hold etoposide |
| AND | |
| Total bilirubin >3 mg/dL or AST >3 times ULN | |

\*\*If enrolled patients on day 6 of therapy have levels of aspartate aminotransferase  $(AST) \ge 2.5 \times UNL$  or alanine aminotransferase  $(ALT) \ge 2.5 \times UNL$  or total bilirubin  $\ge 2 \times ULN$  the administration of GO will be on hold until recovery of total bilirubin to less than or equal to  $2 \times ULN$  and AST and ALT to less than or equal to  $2.5 \times ULN$  prior to each dose. Daily values of LFTs will be obtained. The GO dose can be delayed up to the  $10^{th}$  day after the initiation of therapy due to toxicity or unexpected events (ie infection). Doses of GO will be capped at 4.5 mg. Administration of a FLT3 inhibitor will be prohibited until CR is achieved. The use of a FLT-3 inhibitor is not prohibited after CR has been achieved for patients with FLT3-ITD or FLT-TKD mutations.

| ON STUDY EVALUATION | TIMING |
|---|---|
| History and physical examination | Daily during the hospital stay at UPMC |
| | Shadyside Hospital and then weekly as |
| | outpatient for 4 weeks, and then every 2 |
| | weeks until count recovery |
| CBC with differential | CBC with differential will be performed daily during the inpatient stay and weekly as outpatient until count recovery |

| Complete metabolic panel including LFTs | Complete metabolic panel including liver |
|---|---|
| | function tests (LFTs) will be performed daily |
| | during the admission. After discharge, they |
| | will be followed weekly as outpatient until |
| | count recovery |
| Bone marrow aspiration and biopsy (to | At least 7 days after the completion of |
| evaluate disease status) | treatment |
| Weight | Daily (if clinical possible) while in |
| | hospital and during each visit outpatient |

Bone marrow biopsy, aspirate with flow cytometry studies, cytogenetics and molecular studies will be performed no earlier than 7 days after the completion of treatment. Once hematopoietic recovery has been achieved patients will undergo bone marrow biopsy and/or aspiration for disease evaluation which can be performed in the inpatient or outpatient setting. If the bone marrow is consistent with morphologic complete remission, minimal residual disease testing will be performed with flow cytometry. If on diagnosis the NPM1 mutation was detectable by PCR or next-generation sequencing then NPM1 PCR will be performed as well if morphologic complete remission is achieved If hematopoietic recovery has not been achieved by 5 weeks after the completion of therapy bone marrow biopsy and/or aspiration for disease evaluation will be performed.

| Study Flow Chart | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Screening Period | | Treatment Days | | | | | | Post-treatment | | |
| | Main<br>Study<br>Screening | 1 | 2 | 3 | 4 | 5 | 6 | Daily<br>during<br>Inpatient<br>stay | Follow<br>Up<br>Visits | Survival<br>Follow<br>up <sup>a</sup> |
| Scheduling Window<br>(Days) | -14 to 0 | Can delay each dose<br>up to 3 days. | | | | se | Up to 5 days<br>from the last<br>dose of<br>etoposide/<br>mitoxantrone <sup>b</sup> | | Weekly <sup>c</sup> | |
| Informed Consent | X | | | | | | | | | |
| Inclusion/Exclusion<br>Criteria | Х | | | | | | | | | |

| Medication<br>Review <sup>d</sup> | Х | х | х | х | х | Х | Х | Х | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Trial Treatment Administration | | Х | Х | Х | Х | Х | Х | | | |
| Post-study<br>anticancer therapy<br>status | | | | | | | | | | Х |
| Survival Status | | | | | | | | | | Χ |
| Review Adverse<br>Events | X (from 1st induction therapy) | Х | Х | Х | х | х | Х | Х | х | |
| Full Physical<br>Examination | Х | | | | | | | | Х | |
| Directed Physical<br>Examination | | Х | Х | Х | Х | Х | Х | Х | | |
| Vital Signs and<br>Weight | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| ECOG<br>Performance Status | Х | Х | х | Х | x | Х | × | X | x | |
| Urine or Serum β-<br>HCG | Х | | | | | | | | | |
| PT/INR and aPTT | Xe | | | | | | | | | |
| CBC with differential | Xe | Х | Х | Х | Х | Х | Х | Х | Xf | |
| Comprehensive<br>Serum<br>Chemistry Panel <sup>9</sup> | Хe | Х | х | х | х | х | Х | X | Xf | |
| Magnesium,<br>Phosphorus,<br>Uric Acid, LDH | Xe | Х | х | х | х | х | Х | х | | |
| Urinalysis | Xe | | | | | | | | | |
| Chest Radiograph | Xe | | | | | | | | | |
| Echocardiogram | Xh | | | | | | | | | |
| EKG | Xe | | | | | | | | | |
| Bone Marrow<br>Biopsy | Xi | | | | | | | | Χi | |
| Archival or Newly | Х | | | | | | | | | |
| Obtained Tissue<br>Collection | | | | | | | | | | |

<sup>&</sup>lt;sup>a</sup> Survival will be assessed daily during inpatient stays and then in the follow up visits. After the assessment of the recovery marrow or the marrow after 5 weeks from the completion of therapy patients will be followed remotely from chart review to evaluate the disease-free survival and overall survival. If information cannot be obtained from the chart, patients may be contacted by telephone. <sup>b</sup> Administration of a FLT3 inhibitor will be prohibited until CR is achieved. The use of a FLT-3 inhibitor is not prohibited after CR has been achieved for patients with FLT3-ITD or FLT-TKD mutations.

c After discharge the patient will be followed weekly for 4 weeks and then every 2 weeks until count

recovery (defined as ANC  $\geq$  1000 with or without PLT  $\geq$  100,000). If patients develop grade 3 or 4 nonhematologic toxicity during their treatment they will be followed weekly after discharge until resolution of toxicity or improvement to grade 2 or less. There is  $\pm$  4 days window for each visit. <sup>d</sup> Medication review will be performed from the day of screening until the day of discharge. <sup>e</sup> All screening laboratory assessment must occur within 14 days after consent is signed. <sup>f</sup> After discharge, CBC with differential and complete metabolic panel will be obtained weekly until count recovery (defined as ANC  $\geq$  1000 with or without PLT  $\geq$  100,000). <sup>g</sup> Includes Na, K, Cl, HCO3, BUN, Cr, glucose, Ca, total protein, albumin, total bilirubin, AST, ALT, alkaline phosphatase. <sup>h</sup> Transthoracic Echocardiogram must be performed after the administration of 7 days of cytarabine with 3 days of idarubicin and before the first day of the study treatment. <sup>i</sup> Bone marrow with persistent disease as described in eligibility criteria section and CD33

expression in ≥ 30% leukemic blasts on the bone marrow. <sup>j</sup> Bone marrow biopsy and/or aspirate will be performed no earlier than 7 days after the therapy completion to evaluate disease response. Bone marrow biopsy/aspiration to test for remission once hematopoietic recovery has been achieved will be performed in the inpatient or outpatient setting. If hematopoietic recovery has not been achieved by 5 weeks after the completion of therapy bone marrow biopsy/aspiration for disease evaluation will be performed. If the recovery bone marrow is consistent with morphologic complete remission, minimal residual disease testing will be performed with flow cytometry. If at AML diagnosis the NPM1 mutation was detectable by PCR or next generation sequencing then NPM1 PCR will be performed as well. <sup>k</sup> Blood will be collected prior to the initiation of therapy with mitoxantrone and etoposide, prior to the initiation of therapy with GO, after the administration of GO and weekly while in the hospital. Blood and bone marrow aspirate will be collected at the time of bone marrow evaluation following hematopoietic recovery or prolonged cytopenias.

# **APPENDIX I**

**Performance Status Criteria** 

| ECOG Performance Status Scale | |
|---|---|
| Grade | Descriptions |
| 0 | Normal activity. Fully active, able to carry on all pre-disease performance without restriction. |
| 1 | Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work). |
| 2 | In bed <50% of the time. Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours. |
| 3 | In bed >50% of the time. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours. |
| 4 | 100% bedridden. Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair. |
| 5 | Dead. |

# **APPENDIX II**

# RESPONSE CRITERIA FOR ACUTE LEUKEMIA

# Morphologic leukemia-free state

Bone marrow < 5% blasts in an aspirate with spicules

No blasts with Auer rods or persistence of extramedullary disease Absolute neutrophil count < 1000/mcL AND platelets <100,000/mcL

#### Complete remission

Bone marrow < 5% blasts in an aspirate with spicules Absolute neutrophil count > 1000/mcL

Platelets ≥100,000/mcL

No residual evidence of extramedullary disease

Morphologic CR - patient independent of transfusions

Cytogenetic CR - cytogenetics normal (in those with previously abnormal cytogenetics)

Molecular CR - molecular studies negative

## Complete remission with incomplete hematologic recovery

Bone marrow < 5% blasts in an aspirate with spicules

No residual evidence of extramedullary disease

Absolute neutrophil count > 1000/mcL or platelets ≥100,000/mcL

No residual evidence of extramedullary disease

#### Partial remission

Decrease of at least 50% in the percentage of blasts to 5 to 25% in the bone marrow Patients failing to achieve a complete remission are considered treatment failures

#### Relapse

Relapse following complete remission is defined as reappearance of leukemic blasts in the peripheral blood or the finding of more than 5% blasts in the bone marrow, not attributable to another cause (eg, bone marrow regeneration after consolidation therapy)

Cheson BD, Bennett JM, Kopecky KJ et al. J Clin Oncol 2003;21 (24):4642-4649

#### 9. DRUG INFORMATION

**Gemtuzumab Ozogamicin** 

**Other Names:** Mylotarg

Classification: Antibody-drug conjugate

**Mechanism of Action:** Antibody-drug conjugate to CD33 antigen. Binding results in internalization of the antibody-antigen complex. Following internalization, the calicheamicin derivative is released inside the myeloid cell. The calicheamicin derivative binds to DNA resulting in double strand breaks and cell death. Pluripotent stem cells and

nonhematopoietic cells are not affected.

Storage and Stability: GO is supplied as a sterile, pyrogen-free, unpreserved, white lyophilized powder in amber glass vials. The unopened vials of GO should be stored at

2 - 8° C (refrigerated) and protected from light and should be used within 8 hours of

reconstitution. GO is light sensitive and should be reconstituted, prepared, and

administered under protection from direct/indirect sunlight and Ultraviolet (UV) light.

**Dose Specifics:** GO will be administered at 3 mg/m<sup>2</sup> (cap at 4.5mg) on day 6. BSA will be

calculated based on actual body weight.

**Preparation**: GO is light sensitive and must be protected from direct and indirect sunlight

and unshielded fluorescent light during the preparation and administration of the infusion.

ALL PREPARATION SHOULD BE DONE IN A BIOLOGIC SAFETY HOOD WITH

FLUORESCENT LIGHT OFF. Prior to reconstitution, allow vials to come to room

temperature for approximately 5 minutes. Reconstitute the contents of each vial with 5

mL sterile water for injection, USP, using sterile syringes. Gently swirl each vial. The final

concentration is 1 mg/mL. Use reconstituted solution immediately or after being

refrigerated at 2-8°C for up to 1 hour. Protect reconstituted solution from light. Do not

freeze reconstituted solution. Dilute the desired volume of GO into a 50-milliliter

32

intravenous bag of 0.9% sodium chloride injection or other appropriate volume of 0.9% sodium chloride to make a final GO concentration between 0.075 mg/ml to 0.234 mg/mL. Gently invert the infusion container to mix the diluted solution. Do not shake. Following dilution with 0.9% sodium chloride injection, GO solution should be infused immediately. If not used immediately, store at room temperature (15–25°C; 59–77°F) for up to 6 hours, which includes the 2-hour infusion time and 1-hour, if needed, to allow the refrigerated diluted solution to equilibrate to room temperature. The diluted solution can be refrigerated at 2–8°C (36–46°F) for up to 12 hours which includes up to 1-hour in the vial post-reconstitution.

**Route of Administration:** GO is administered as a 2 hour IV infusion. A 0.2-micron polyethersulfone filter is required on the IV line. The IV bag must be protected from light using a light-blocking cover during infusion. The infusion line does not need to be protected from light.

**Compatibilities:** No information; infuse via separate line.

Availability: Commercially available

#### Side Effects:

**Common** (occurs in more than 10% of people - more than 10 out of 100 people): fever (79%), infection (42%), increased AST (40%), sepsis (32%), bleeding (23%), nausea and vomiting (21%), constipation (21%), mucositis (21%), headache (19%), increased ALT (16%), rash (16%)

*Infrequent* (occurs in 1% to 10% of people - from 1 to 10 out of 100 people): pneumonia (7%), bleeding (7%), hyperbilirubinemia (7%), mucositis (4%), pain (4%), diarrhea (2%), headaches (2%), tachycardia (2%), lung edema (2%)

Rare (occurs in <1% of people, mainly identified in post-marketing surveillance):

neutropenic colitis, interstitial pneumonia, hemorrhagic cystitis

Nursing Implications: Patients should be premedicated prior to administration of GO

with methylprednisolone 1 mg/kg IV, diphenhydramine 50 mg IV or PO and

acetaminophen 650 mg PO 30 minutes prior to start of the infusion. Additional doses of

acetaminophen and diphenhydramine may be administered every 4 hours after the initial

pretreatment dose. Repeat with the same dose of methylprednisolone for any sign of an

infusion reaction, such as fever, chills, hypotension, or dyspnea during the infusion or

within 4 hours afterwards.

During and after the infusion patients will be monitored with vital signs recorded every

30 minutes during the infusion and for 1 hour after completion of the infusion.

GO should be administered in a setting where appropriate medical support, including life

support equipment, is available in case of an unexpected adverse event.

**Etoposide** 

Other Names: Toposar

Classification: Podophyllotoxin Derivative

**Mechanism of Action:** Etoposide has been shown to delay transit of cells through the S

phase and arrest cells in late S or early G<sub>2</sub> phase. The drug may inhibit mitochondrial

transport at the NADH dehydrogenase level or inhibit uptake of nucleosides into HeLa cells.

It is a topoisomerase II inhibitor and appears to cause DNA strand breaks. Etoposide does

not inhibit microtubular assembly.

Storage and Stability: Unopened vials of etoposide are stable for 24 months at room

temperature (25 degrees Celsius). Vials of etoposide are stable at room temperature for 96

34

hours when diluted to concentrations of 0.2 milligrams/milliliter (mg/mL); stability is 24 hours with concentrations of 0.4 mg/mL at room temperature. The manufacturer does not recommend that etoposide be administered at concentrations greater than 0.4 mg/mL because time to precipitation is highly unpredictable and precipitate formation has been reported to occur earlier than the utility times listed above. Etoposide 20 mg/ml is stable in a plastic syringe for 5 days when stored at room temperature under fluorescent light.

**Dose Specifics:** Patients will receive etoposide 100 mg/m² administered intravenously in 500 ml of 0.9% sodium chloride over 2 hours on days 1-5 (for patients who have elevated total bilrirubin, AST or reduced creatinine clearance during the etoposide infusion see treatment schema for dose modification of the etoposide). BSA will be calculated based on actual body weight.

**Preparation:** Etoposide Injection must be diluted prior to use with either 5% Dextrose Injection, or 0.9% Sodium Chloride Injection, to give a final concentration of 0.2 to 0.4 mg/mL. If solutions are prepared at concentrations above 0.4 mg/mL, precipitation may occur. Parenteral drug products should be inspected visually for particulate matter and discoloration prior to administration whenever solution and container permit.

**Route of Administration:** Etoposide should be given as a diluted solution via the IV route.

**Compatibilities:** Variable stability (consult detailed reference) in D<sub>5</sub>W, LR, NS.Y-site administration: Compatible: Allopurinol, amifostine, aztreonam, cladribine, doxorubicin liposome, fludarabine, gemcitabine, granisetron, melphalan, ondansetron, paclitaxel, piperacillin/tazobactam, sargramostim, sodium bicarbonate, teniposide, thiotepa, topotecan, vinorelbine. Incompatible: Cefepime, filgrastim, idarubicin.

**Compatibility when admixed:** Compatible: Carboplatin, cisplatin, with cyclophosphamide, cisplatin with floxuridine, cytarabine, cytarabine with daunorubicin, floxuridine, fluorouracil, hydroxyzine, ifosfamide, ifosfamide with carboplatin, ifosfamide

with cisplatin, ondansetron. Variable (consult detailed reference): Cisplatin with mannitol

and potassium chloride, doxorubicin with vincristine.

**Availability:** Commercially available

Side Effects:

**Common** (occurs in more than 10% of people - more than 10 out of 100 people):

Alopecia (8% to 66%), ovarian failure (38%), Nausea/vomiting (31% to 43%), anorexia

(10% to 13%), diarrhea (1% to 13%), leukopenia (60 to 91%), thrombocytopenia (22%)

to 41%), anemia (up to 33%), mucositis

**Infrequent** (occurs in 1% to 10% of people - from 1 to 10 out of 100 people):

Hypotension (1% to 2%), stomatitis (1% to 6%), abdominal pain (up to 2%), hepatic

toxicity (up to 3%), peripheral neuropathy (1% to 2%), anaphylactic-like reaction (IV

infusion 1% to 2%)

**Rare** (occurs in fewer than 1% of people – fewer than 1 out of 100 people):

Congestive heart failure, hyperpigmentation, rash, radiation-recall reaction,

Stevens Johnson Syndrome, pruritus, toxic epidermal necrolysis, cyanosis, optic neuritis,

transient blindness, diaphoresis, interstitial pneumonitis, pulmonary fibrosis, metabolic

acidosis, thrombophlebitis, extravasation

Nursing Implications: For IV use only; may cause severe local tissue damage if

extravasation occurs. Do not administer intrathecally; may cause serious and permanent

neurologic damage. Should be administered under the supervision of an experienced

cancer chemotherapy physician.

Mitoxantrone

36

Other Names: Dihydroxyanthracenedione, DHAD

Classification: Anthracenedione

**Mechanism of Action:** Analogue of the anthracyclines, mitoxantrone intercalates DNA;

binds to nucleic acids and inhibits DNA and RNA synthesis by template disordering and

steric obstruction; replication is decreased by binding to DNA topoisomerase II and seems

to inhibit the incorporation of uridine into RNA and thymidine into DNA; active throughout

entire cell cycle

Storage and Stability: Intact vials should be stored between 15 and 25 degrees Celsius

(59 and 77 degrees Fahrenheit). DO NOT FREEZE. After penetration of the stopper, store

the remaining solution of undiluted mitoxantrone for no longer than 7 days between 15 to

25 degrees Celsius (59 to 77 degrees Fahrenheit) or for no longer than 14 days under

refrigeration (2 to 8 degrees Celsius or 36 to 46 degrees Fahrenheit). Mitoxantronemust

be further diluted for infusion.

**Dose Specifics:** Patients will receive mitoxantrone 10mg/m<sup>2</sup> administered IVPB in 50ml

0.9% sodium chloride over 15 minutes on days 1-5. (Refer to Treatment Plan of Phase I

and II sections). BSA will be calculated based on actual body weight.

Preparation: MITOXANTRONE CONCENTRATE MUST BE DILUTED PRIOR TO USE.

Dilute the dose with at least 50 milliliters (mL) of 0.9% sodium chloride or 5% dextrose in

water. Dilution in volumes greater than 50 mL may be done in 5% dextrose in water, 0.9%

sodium chloride, or dextrose 5% with 0.9% sodium chloride. Parenteral drug products

should be inspected visually for particulate matter and discoloration prior to administration

whenever solution and container permit.

Route of Administration: Mitoxantrone should be given as a diluted solution via the IV

route.

37

**Compatibilities:** Stable in D<sub>5</sub>NS, D<sub>5</sub>W, NS Y-site administration: Compatible: Allopurinol, amifostine, cladribine, etoposide phosphate, filgrastim, fludarabine, gatifloxacin, gemcitabine, granisetron, linezolid, melphalan, ondansetron, sargramostim, teniposide, thiotepa, vinorelbine. Incompatible: Amphotericin B cholesteryl sulfate complex, aztreonam, cefepime, doxorubicin liposome, paclitaxel, piperacillin/tazobactam, propofol.

**Compatibility when admixed:** Compatible: Cyclophosphamide, cytarabine, fluorouracil, hydrocortisone sodium succinate, potassium chloride. Incompatible: Heparin. Variable (consult detailed reference): Hydrocortisone sodium phosphate.

Availability: Commercially available

#### Side Effects:

Common (occurs in more than 10% of people - more than 10 out of 100 people): Arrhythmia (3% to 18%), ECG changes (11%), fatigue (up to 39%), fever (6% to 78%), headache (6% to 13%), alopecia (20% to 61%), nail bed changes (11%), amenorrhea (28% to 53%), menstrual disorder (26% to 61%), hyperglycemia (10% to 31%), abdominal pain (9% to 15%), anorexia (22% to 25%), nausea (26% to 76%), constipation (10% to 16%), diarrhea (14% to 47%), GI bleeding (2% to 16%), mucositis (10% to 29%), stomatitis (8% to 29%), vomiting (6% to 11%), urinary tract infection (7% to 32%), neutropenia (79% to 100%), leukopenia (9% to 100%), lymphopenia (72% to 95%), anemia (5% to 75%), thrombocytopenia (33% to 39%), petechiae/bruising (6% to 11%), alkaline phosphatase increased (37%), transaminases increased (5% to 20%), creatinine increased (13%), hematuria (11%), dyspnea (6% to 18%), upper respiratory tract infection (7% to 53%), fungal infection (9% to 15%), infection (4% - 18%), sepsis (31% to 34%)

**Infrequent** (occurs in 1% to 10% of people - from 1 to 10 out of 100 people): LVEF decreased (≤5%), CHF (2% - 5%), depression (5%), seizure (2% - 4%), hypocalcemia

(10%), hypokalemia (7% - 10%), hyponatremia (9%), menorrhagia (7%),impotence (7%), jaundice (3% to 7%), myalgia (5%), arthralgia (5%), conjunctivitis (5%), blurred vision (3%), renal failure (8%), proteinuria (6%), rhinitis (10%), pneumonia (9%), sinusitis (6%), diaphoresis (9%)

**Rare** (occurs in fewer than 1% of people – fewer than 1 out of 100 people): Blue skin discoloration, rash, interstitial pneumonitis, hypersensitivity, extravasation

May cause myocardial toxicity and potentially-fatal congestive heart failure (CHF); risk increases with cumulative dosing. Predisposing factors for mitoxantrone-induced cardiotoxicity include prior anthracycline therapy, prior cardiovascular disease, concomitant use of cardiotoxic drugs, and mediastinal/pericardial irradiation. Not recommended for use when left ventricular ejection fraction (LVEF) <50%.

**Nursing implications:** For IV use only; may cause severe local tissue damage if extravasation occurs. Do not administer intrathecally; may cause serious and permanent neurologic damage. May cause urine, saliva, tears, and sweat to turn blue-green for 24 hours post infusion. Whites of eyes may have blue-green tinge. Has been associated with the development of secondary acute myelogenous leukemia and myelodysplasia. Should be administered under the supervision of an experienced cancer chemotherapy physician.

#### 10. REFERENCES

#### References

- 1. Dohner H, Weisdorf DJ, Bloomfield CD. Acute Myeloid Leukemia. *N Engl J Med*. 2015;373(12):1136-1152.
- 2. Rowe JM, Tallman MS. How I treat acute myeloid leukemia. *Blood*. 2010;116(17):31473156.
- 3. Kolitz JE. Current therapeutic strategies for acute myeloid leukaemia. *Br J Haematol*. 2006;134(6):555-572.
- 4. Orlowski RJ, Mangan JK, Luger SM. Approach to patients with primary refractory acute myeloid leukemia. *Curr Opin Hematol.* 2015;22(2):97-107.

- 5. Hamann PR, Hinman LM, Hollander I, et al. Gemtuzumab ozogamicin, a potent and selective anti-CD33 antibody-calicheamicin conjugate for treatment of acute myeloid leukemia. *Bioconjug Chem.* 2002;13(1):47-58.
- 6. Yamauchi T, Matsuda Y, Tasaki T, et al. Induction of DNA strand breaks is critical to predict the cytotoxicity of gemtuzumab ozogamicin against leukemic cells. *Cancer Sci.* 2012;103(9):1722-1729.
- 7. Khan N, Hills RK, Virgo P, et al. Expression of CD33 is a predictive factor for effect of gemtuzumab ozogamicin at different doses in adult acute myeloid leukaemia. *Leukemia*. 2017;31(5):1059-1068.
- 8. Sievers EL, Larson RA, Stadtmauer EA, et al. Efficacy and safety of gemtuzumab ozogamicin in patients with CD33-positive acute myeloid leukemia in first relapse. *J Clin Oncol*. 2001;19(13):3244-3254.
- 9. Bross PF, Beitz J, Chen G, et al. Approval summary: gemtuzumab ozogamicin in relapsed acute myeloid leukemia. *Clin Cancer Res.* 2001;7(6):1490-1496.
- 10. Petersdorf SH, Kopecky KJ, Slovak M, et al. A phase 3 study of gemtuzumab ozogamicin during induction and postconsolidation therapy in younger patients with acute myeloid leukemia. *Blood*. 2013;121(24):4854-4860.
- 11. Castaigne S, Pautas C, Terre C, et al. Effect of gemtuzumab ozogamicin on survival of adult patients with de-novo acute myeloid leukaemia (ALFA-0701): a randomised, openlabel, phase 3 study. *Lancet*. 2012;379(9825):1508-1516.
- 12. Amadori S, Suciu S, Selleslag D, et al. Gemtuzumab Ozogamicin Versus Best Supportive Care in Older Patients With Newly Diagnosed Acute Myeloid Leukemia Unsuitable for Intensive Chemotherapy: Results of the Randomized Phase III EORTC-GIMEMA AML19 Trial. *J Clin Oncol.* 2016;34(9):972-979.
- 13. Burnett A, Cavenagh J, Russell N, et al. Defining the dose of gemtuzumab ozogamicin in combination with induction chemotherapy in acute myeloid leukemia: a comparison of 3 mg/m2 with 6 mg/m2 in the NCRI AML17 Trial. *Haematologica*. 2016;101(6):724-731.
- 14. Larson RA, Sievers EL, Stadtmauer EA, et al. Final report of the efficacy and safety of gemtuzumab ozogamicin (Mylotarg) in patients with CD33-positive acute myeloid leukemia in first recurrence. *Cancer*. 2005;104(7):1442-1452.
- 15. Magwood-Golston JS, Kessler S, Bennett CL. Evaluation of gemtuzumab ozogamycin associated sinusoidal obstructive syndrome: Findings from an academic pharmacovigilance program review and a pharmaceutical sponsored registry. *Leuk Res.* 2016;44:61-64.
- 16. Tallman MS, McDonald GB, DeLeve LD, et al. Incidence of sinusoidal obstruction syndrome following Mylotarg (gemtuzumab ozogamicin): a prospective observational study of 482 patients in routine clinical practice. *Int J Hematol.* 2013;97(4):456-464.
- 17. Wadleigh M, Richardson PG, Zahrieh D, et al. Prior gemtuzumab ozogamicin exposure significantly increases the risk of veno-occlusive disease in patients who undergo myeloablative allogeneic stem cell transplantation. *Blood.* 2003;102(5):1578-1582.
- 18. Battipaglia G, Labopin M, Candoni A, et al. Risk of sinusoidal obstruction syndrome in allogeneic stem cell transplantation after prior gemtuzumab ozogamicin treatment: a retrospective study from the Acute Leukemia Working Party of the EBMT. *Bone Marrow Transplant*. 2017;52(4):592-599.
- 19. Burnett AK, Hills RK, Hunter AE, et al. The addition of gemtuzumab ozogamicin to lowdose Ara-C improves remission rate but does not significantly prolong survival in

- older patients with acute myeloid leukaemia: results from the LRF AML14 and NCRI AML16 pick-a-winner comparison. *Leukemia*. 2013;27(1):75-81.
- 20. Burnett AK, Hills RK, Milligan D, et al. Identification of patients with acute myeloblastic leukemia who benefit from the addition of gemtuzumab ozogamicin: results of the MRC AML15 trial. *J Clin Oncol.* 2011;29(4):369-377.
- 21. Castaigne S, Pautas C, Terré C, et al. Final Analysis of the ALFA 0701 Study. *Blood*. 2014;124(21):376-376.
- 22. Burnett AK, Russell NH, Hills RK, et al. Addition of gemtuzumab ozogamicin to induction chemotherapy improves survival in older patients with acute myeloid leukemia. *J Clin Oncol.* 2012;30(32):3924-3931.
- 23. Amadori S, Suciu S, Stasi R, et al. Sequential combination of gemtuzumab ozogamicin and standard chemotherapy in older patients with newly diagnosed acute myeloid leukemia: results of a randomized phase III trial by the EORTC and GIMEMA consortium (AML-17). *J Clin Oncol*. 2013;31(35):4424-4430.
- 24. Lowenberg B, Beck J, Graux C, et al. Gemtuzumab ozogamicin as postremission treatment in AML at 60 years of age or more: results of a multicenter phase 3 study. *Blood*. 2010;115(13):2586-2591.
- 25. McHayleh W, Sehgal R, Redner RL, et al. Mitoxantrone and etoposide in patients with newly diagnosed acute myeloid leukemia with persistent leukemia after a course of therapy with cytarabine and idarubicin. *Leuk Lymphoma*. 2009;50(11):1848-1853.
- 26. Boyiadzis M, Redner RL, Raptis A, Hou JZ, Agha M, Foon KA. Gemtuzumab ozogamicin, mitoxantrone, and etoposide in newly diagnosed acute myeloid leukemia patients with persistent leukemia after a course of induction therapy. *Ann Hematol*. 2011;90(6):733-735.
- 27. van der Velden VH, Boeckx N, Jedema I, et al. High CD33-antigen loads in peripheral blood limit the efficacy of gemtuzumab ozogamicin (Mylotarg) treatment in acute myeloid leukemia patients. *Leukemia*. 2004;18(5):983-988.
- 28. Boyiadzis M, Whiteside TL. Information transfer by exosomes: A new frontier in hematologic malignancies. *Blood Rev.* 2015;29(5):281-290.
- 29. Boyiadzis M, Whiteside TL. The emerging roles of tumor-derived exosomes in hematological malignancies. *Leukemia*. 2017;31(6):1259-1268.
- 30. Aung T, Chapuy B, Vogel D, et al. Exosomal evasion of humoral immunotherapy in aggressive B-cell lymphoma modulated by ATP-binding cassette transporter A3. *Proc Natl Acad Sci U S A*. 2011;108(37):15336-15341.
- 31. Oksvold MP, Kullmann A, Forfang L, et al. Expression of B-cell surface antigens in subpopulations of exosomes released from B-cell lymphoma cells. *Clin Ther*. 2014;36(6):847-862 e841.
- 32. Ciravolo V, Huber V, Ghedini GC, et al. Potential role of HER2-overexpressing exosomes in countering trastuzumab-based therapy. *J Cell Physiol*. 2012;227(2):658-667.
- 33. Hong CS, Funk S, Muller L, Boyiadzis M, Whiteside TL. Isolation of biologically active and morphologically intact exosomes from plasma of patients with cancer. *J Extracell Vesicles*. 2016;5:29289.